CLINICAL TRIAL: NCT02866929
Title: Molecular Evaluation of Inflammatory and Bone Remodeling Markers in Gingival Crevicular Fluid After Selective Alveolar Decortication
Brief Title: A Biotype Enhancing Strategy For The Patient Undergoing Accelerated Orthodontics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CES University (Other)
Collaborators: University of Michigan (Other); Universidad del Valle, Colombia (Other)
Responsible Party: Principal Investigator, Maria Antonia Alvarez, Researcher, CES University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ODCES001
Record Dates: First submitted 2016-07-06; First posted 2016-08-15 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Class I Malocclusion; Other Periodontal Diseases; Thin Gingival Biotype
Keywords: orthodontics; periodontics; piezosurgery; accelerated orthodontics; Surgically Accelerated Orthodontic Treatment
MeSH Terms: conditions — Malocclusion, Angle Class I | interventions — Cerebral Decortication; Orthodontics; Mucograft

ARMS (4):
- Conventional orthodontic treatment (Active Comparator): Patients that will receive conventional orthodontics
  Interventions: Device: Orthodontics
- Orthodontics with decortication (Experimental): Patients that will receive orthodontic treatment with selective alveolar decortication
  Interventions: Procedure: Decortication; Device: Orthodontics
- Orthodontics decortication and Mucograft (Experimental): Orthodontic treatment, selective alveolar decortication and Mucograft® on the mandibular anterior segment
  Interventions: Procedure: Decortication; Device: Orthodontics; Drug: Mucograft
- Orthodontics and Mucograft® (Experimental): Patients that will receive orthodontic treatment and Mucograft® on the mandibular anterior segment
  Interventions: Device: Orthodontics; Drug: Mucograft

INTERVENTIONS:
Procedure: Decortication — Under local anesthesia, vertical and inter-radicular gingival incisions will be performed on the vestibular of the maxillary and mandibular arch, starting 2-3 mm below the interdental papilla and with sufficient depth to the periosteum to allow the scalpel to reach the alveolar bone. These incisions will be kept as small as possible; then, through them, using a piezoelectric scalpel (piezotome), several bone cuts will be performed. These cuts will have sufficient depth for drilling the cortical alveoli.
  Arms: Orthodontics decortication and Mucograft; Orthodontics with decortication
Device: Orthodontics — Self-ligation brackets in upper and lower teeth
Drug: Mucograft — Porcine naturally cross-linked collagen matrix
  Arms: Orthodontics and Mucograft®; Orthodontics decortication and Mucograft

SUMMARY:
Numerous treatment protocols geared towards accelerating orthodontic treatment have emerged in the past few years as an appealing alternative for patients and practitioners. In the context of a thin biotype, these approaches pose a burden that could precipitate periodontal detrimental changes. Therefore, case selection and the implementation of periodontal biotype enhancing strategies become a relevant consideration to ensure long-term successful treatment outcomes. This study focuses on the biological and clinical value of the use of a porcine naturally cross-linked collagen matrix known as Mucograft®. Within the scope of Surgically Accelerated Orthodontic Treatment (SAOT) the structural and material features of Mucograft® provide: 1) A protective effect to the thin biotype upon rapid orthodontic protusive/proinclination movements and 2) Mucograft® enhances the therapeutic window effect that supports an increase on tooth movement rate. The designs of this randomized controlled clinical trial includes a cohort of 40 subjects distributed on the following groups I) Ortho tx, II) Ortho tx + Decortication, III) Ortho tx + Decortication + Mucograft®, and IV) Ortho tx + Mucograft®. Comparing clinical, tomographic and digital impression derived measurements will capture the clinical phenotype; while the biologic phenotype will be derived from evaluating crevicular fluid levels of tooth movement mediators such as Interleukin 1-β and Interleukin-1RA. The significance and innovative value of this proposal stems from the use of Mucograft® as an ideal collagen-based biotype enhancer when performed along with the corticotomy. This approach could prove to be effective to further increase the therapeutic window that allows accelerating orthodontic treatment and, at the same time, could decrease the recession risk in movements of proclination of antero-inferior incisors. Besides, the use of a collagen scaffold alone could potentially trigger a comparable orthodontic acceleratory outcome that could be evaluated as an alternative to decortication.

ELIGIBILITY:
Inclusion Criteria:

* Angle's class I malocclusion
* Little's grade II or III dental crowding
* Periodontally stable patients
* Patients with no more than 2 mm of keratinized gingiva in at least two sites of the antero-inferior region

Exclusion Criteria:

Patient with presence of marginal tissue recessions on inferior incisors

* Patients with a metabolic or neoplastic alteration
* History of orthopedic surgery in the last 6 months
* History of fractures in the last 6 months
* History of bisphosphonates use
* Patient with systemic compromise

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Volumetric changes of soft tissue in relation to underlying bone using 3D reconstruction models. | 2 years

SECONDARY OUTCOMES:
Levels of pro-inflammatory cytokines, derived from gingival crevicular fluid, associated with tooth movement. | 4 weeks
Determining the safety and efficacy of the Mucograft by comparing periodontal stability at baseline and post-treatment, taking clinical periodontal measures. | 2 years
Measuring tooth movement rate based on changes of tooth alignment using superimposition of digital impressions of the mandibular anterior region of interest. | 2 years